CLINICAL TRIAL: NCT00455208
Title: Study Evaluating Cura-100 in Rheumatoid Arthritis and Osteoarthritis
Brief Title: A Study Evaluating the Safety and Efficacy of Cura-100 in Subjects With Rheumatoid Arthritis and Osteoarthritis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cura Biotech LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CURA-07-10
Record Dates: First submitted 2007-03-30; First posted 2007-04-03 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2007-03

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cura-100

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of Cura-100 in treating rheumatoid arthritis and osteoarthritis.

DETAILED DESCRIPTION:
This is the Phase I/II trial, which monitors both safety and efficacy of Cura-100 in subjects with rheumatoid arthritis and osteoarthritis at one clinical study center. The open-label clinical study will be used in the study. The study is expected to last for one and a half year after it has been officially started, which include recruitment, study treatment and follow-ups. The healthy volunteers are also included to study the safety of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of rheumatoid arthritis and osteoarthritis at active stage
* Able and willing to comply with study visits and procedures specified in this protocol for at least six months period
* Able to understand and willing to sign and date the written informed consent form prior to admission of the study
* Able and willing to provide adequate information for locator purposes
* Able and willing to provide self evaluation information and diagnostic report of arthritis as required for efficacy evaluation

Exclusion Criteria:

* Pregnant women
* Over-weighted
* Hypertension, or diabetes, or a history of cardiovascular disease or kidney disease, or serious skin allergy or other concurrent clinically significant illness or medical condition (other than arthritis) which, in the viewpoint of the study doctor, may put the subject at a possible risk for participation
* Patients used biologic modifier therapy or currently taking immunosuppressive agents might be excluded
* Unable to spend 3 hours for treatment at the study center

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-05; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is remission of rheumatoid arthritis and osteoarthritis, which will be measured with ACR criteria.

SECONDARY OUTCOMES:
The secondary outcome is the reduction in signs and symptoms of rheumatoid arthritis and osteoarthritis for a continuous three or six month period, measured with ACR20 and the change from baseline in HAQ.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Zhang, Study Director — Cura Biotech LLC
Locations (1):
- Cura Biotech LLC, Sunnyvale, California, United States